CLINICAL TRIAL: NCT01287897
Title: A Double-blind, Randomized, Placebo-controlled, Dose-ranging Study To Evaluate The Efficacy And Safety Of Pf-04236921 In Subjects With Crohn's Disease Who Are Anti-tnf Inadequate Responders (Andante)
Brief Title: A Study To Assess The Efficacy And Safety Of PF-04236921 In Subjects With Crohn's Disease Who Failed Anti-TNF Therapy
Acronym: ANDANTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B0151003; 2010-023034-23 (EudraCT Number); ANDANTE (Other: Alias Study Number)
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Results first posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; safety; efficacy; pharmacokinetics; pharmacodynamics; Crohn's Disease Activity Index (CDAI)
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo- SC injection (Placebo Comparator)
  Interventions: Drug: PF-04236921 SC injection
- Drug Dose level 1 - SC injection (Experimental)
  Interventions: Drug: PF-04236921 SC injection
- Drug Dose level 2 - SC injection (Experimental)
  Interventions: Drug: PF-04236921 SC injection

INTERVENTIONS:
Drug: PF-04236921 SC injection — Placebo delivered SC, 2 doses separated by 4 weeks
  Arms: Placebo- SC injection
Drug: PF-04236921 SC injection — Drug dose level 1 delivered SC, 2 doses separated by 4 weeks
  Arms: Drug Dose level 1 - SC injection
Drug: PF-04236921 SC injection — Drug dose level 2 delivered SC, 2 doses separated by 4 weeks
  Arms: Drug Dose level 2 - SC injection

SUMMARY:
This is a proof of concept study to determine the efficacy and safety of a monoclonal antibody with three doses versus placebo. Subjects will be randomized to a treatment and the dose will be delivered subcutaneously twice, 4 weeks apart. All subjects will have moderate to severe refractory Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have failed or are intolerant to anti TNFs
* hsCRP greater or equal to 5.0 mg/L
* Ulcerations demonstrated by colonoscopy as defined by SES CD assessment performed within 8 weeks of study entry (screening) and able to retrospectively complete the SES-CD or colonoscopy performed during screening

Exclusion Criteria:

* Pregnant or breastfeeding women
* Crohn's Disease with active fistulae or abscess
* History of diverticulitis or symptomatic diverticulosis
* Abnormality in hematology or chemistry profiles at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-02; Primary Completion 2014-09 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (192):
- United States (97):
  - UAB Hospital, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Simon Medical Imaging, Scottsdale, Arizona
  - Digestive Health Research Unit, Scottsdale, Arizona
  - Adobe Clinical Research, Llc, Tucson, Arizona
  - Radiology Ltd, Tucson, Arizona
  - UCSF Endoscopy Unit at Mount Zion, San Francisco, California
  - University of California - San Francisco, San Francisco, California
  - University of California San Francisco at Mount Zion, San Francisco, California
  - Rocky Mountain Clinical Research, LLC, Denver, Colorado
  - Rocky Mountain Gastroenterology Associates, Lakewood, Colorado
  - Rocky Mountain Gastroenterology, Lakewood, Colorado
  - Arapahoe Gastroenterology, PC, Littleton, Colorado
  - Endoscopy Center of Connecticut, LLC, Guilford, Connecticut
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Gastroenterology Associates, Crystal River, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - Suncoast Endoscopy Center, Inverness, Florida
  - Advanced Research Institute, Inc., New Port Richey, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Atlanta Endoscopy Center, Decatur, Georgia
  - Decatur Health Imaging, Decatur, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - GI Diagnostics, Marietta, Georgia
  - Illinois Gastroenterology Group, LLC, Arlington Heights, Illinois
  - The University of Chicago Medical Center (Ucmc), Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - The University of Chicago Medical, Chicago, Illinois
  - The University Of Chicago, Chicago, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Glenbrook Hospital Outpatient Pharmacy, Glenview, Illinois
  - Glenbrook Hospital, Glenview, Illinois
  - Central Indiana Gastroenterology Group, Anderson, Indiana
  - Saint John's Research Institute, Anderson, Indiana
  - University of Kentucky, Lexington, Kentucky
  - University Of Louisville Healthcare Outpatient Center, Louisville, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Digestive Disorders Associates, Annapolis, Maryland
  - Disgestive Disorders Associates, Annapolis, Maryland
  - Investigative Clinical Research, Annapolis, Maryland
  - Maryland Diagnostics & Therapeutic Endo Center, Annapolis, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Prima CARE, PC, Fall River, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - East Valley Endoscopy, Grand Rapids, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Metro Health Hospital Endoscopy Unit, Wyoming, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - St. Joseph Mercy Hospital, Ypsilanti, Michigan
  - Minnesota Gastroenterology, PA, Plymouth, Minnesota
  - Weill Cornell Medical College of Cornell University-Greenberg, New York, New York
  - Weill Cornell Medical College of Cornell University, New York, New York
  - Present Chapman, Steinlauf and Marion, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical College Investigational Pharmacy, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Imaging at New York Presbyterian Hospital, New York, New York
  - Arthur asher Kornbluth, MD PC, New York, New York
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Pharmacy: Wheeler and Stuckey, Inc., Oklahoma City, Oklahoma
  - Colonoscopy and X-rays: OU Physicians Building, Oklahoma City, Oklahoma
  - Hillcrest Medical Center Endoscopy, Tulsa, Oklahoma
  - Hillcrest Medical Center, Tulsa, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Utica Park Clinic X-Ray, Tulsa, Oklahoma
  - Advanced Imaging, Tulsa, Oklahoma
  - Pittsburgh Gastroenterology Associates, Pittsburgh, Pennsylvania
  - Research Protocol Management Specialists, Pittsburgh, Pennsylvania
  - Pharma Resource, East Providence, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Professional Quality Research, Inc., Austin, Texas
  - Diagnostic Clinic of Houston, PA, Houston, Texas
  - Houston Hospital for Specialized Surgery (Endoscopy Only), Houston, Texas
  - Baylor Clinic (Drug Storage), Houston, Texas
  - Baylor College of Medicine - Baylor Medical Center, Houston, Texas
  - Ertan Digestive Disease Center, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - Physicians Endoscopy Center (Colonoscopy), Houston, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - One Step Diagnostic (X-Ray), Sugar Land, Texas
  - Pioneer Research Solutions, Inc. (Admin. Office), Sugar Land, Texas
  - Pioneer Research Solutions, Inc., SugarLand, Texas
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - University Of Utah HSC, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - VCU Medical Investigational Drug Service (IDS), Richmond, Virginia
- Australia (8):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Public Hospital, Kingswood, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Brisbane, Queensland
  - Mater Health Services, South Brisbane, Queensland
  - Eastern Health, Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy
- Belgium (4):
  - University Hospital Leuven, Leuven, Vlaams Brabant
  - CHU Saint-Pierre, Brussels
  - UZ Leuven Pharmacy, Leuven
  - An Spiessens H.-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Brazil (8):
  - Clinica do Coracao Samaritano, Goiânia, Goiás
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda., Goiânia, Goiás
  - Center X Diagnosticos, Goiânia, Goiás
  - Hospital Universitário Fraga Filho da UFRJ, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo, São Paulo
  - Hospital Nossa Senhora das Gracas, Curitiba
- Canada (4):
  - Heritage Medical Research Clinic - University of Calgary, Calgary, Alberta
  - London Health Science Centre - University Hospital, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - McGill University Health Centre - Royal Victoria Hospital, Montreal, Quebec
- Czechia (8):
  - Klinicke centrum ISCARE I.V.F. - gastroenterologie, Prague, Prague
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Medial Pharma s.r.o.,, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Institut klinicke a experimentalni mediciny, Prague
  - IBD Clinical and Research centre, Prague
  - Krajska zdravotni, a.s., Ústí nad Labem
- Denmark (8):
  - Aalborg Sygehus, Aalborg
  - Aarhus Universitetshospital, Aarhus Sygehus Aarhus University Hospital, Aarhus C
  - Rigshospitalet, Copenhagen
  - Gastroenheden, Herlev
  - Kirurgisk Afdeling 0143, Hilleroed
  - Hvidovre Hospital, Hvidovre
  - Afdeling I, Gastroenterologisk Sektion, Koebenhavn NV
  - Medicinsk Afdeling, Gastroenterologisk Sektion, Koege
- France (3):
  - Hopital Huriez, CHRU de Lille, Lille
  - Hopital Saint-Antoine - Service De Gastroenterologie, Paris
  - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (6):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - "Charite - Campus Benjamin Franklin, Berlin
  - Praxis Dr. Howaldt, Hamburg
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Universitaetsklinik Regensburg, Regensburg
- Greece (2):
  - University General Hospital "Attikon", Athens
  - General Hospital of Athens "Evangelismos",1st Gastroenterology Department, Kolonaki Athens
- Hungary (6):
  - Semmelweis Egyetem II. Sz. Belgyogyaszati Klinika, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak./I. Belgyogyaszati-Gasztroenterologiai, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar / I. sz. Belgyogyaszati Klinika, Szeged
  - Clinfan Kft., Szekszárd
- Ireland (6):
  - Beaumont Hospital, Dublin
  - National Virus Reference Laboratory, Dublin
  - Pathology, Haematology and Biochemistry Laboratories, St Vincent's Healthcare Group, Dublin
  - Mater Misericordiae Hospital, Department of Clinical Chemistry and Clinical Haematology, Dublin
  - St. Vincents University Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (9):
  - The Institute Of Gastroenterology & Liver Diseases, Tel Litwinsky, Ramat Gan
  - Institute of Gastroenterology, Haifa
  - The E. Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Dept of Gastroenterology & Hepatology, Kfar Saba
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (8):
  - Casa Sollievo della Sofferenza/Div.Gastroenterologia Endoscopia Digestiva, San Giovanni Rotondo Fg, Foggia
  - Istituto Clinico Humanitas IRCCS, Rozzano, Milano
  - Azienda Ospedaliera - Universita di Padova, Padua, Padova
  - A. Gemelli University Hospital-Department of Medical Sciences - Division of Internal Medicine and, Rome, Province of Rome
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola Malpighi, Bologna
  - Università Campus Biomedico, Roma
  - Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera San Camillo Forlanini, Roma
- New Zealand (4):
  - Shakespeare Specialist Group, Milford, Auckland
  - Christchurch Hospital, Christchurch, Canterbury
  - Department of Gastroenterology Research, Hamilton, Waikato Region
  - P3 Research Limited, Wellington
- Spitalul Clinic Colentina, Bucharest, Sector 2, Romania
- Universitaetsspital Zuerich, Zurich, Switzerland
- United Kingdom (9):
  - Hull and East Yorkshire Hospitals NHS Trust, Hull, East Yorkshire
  - Addenbrooke's Hospital, Department of Gastroenterology, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - Pharmacy Department, Hull
  - Barts and The London NHS Trust, London
  - Royal Free Hospital (Royal Free London NHS Foundation Trust), London
  - Royal Victoria Hospital, Newcastle upon Tyne
  - New Cross Hospital, Wolverhampton
  - Newcross Hospital-The Royal Wolverhampton Hospitals NHS Trust, Wolverhampton

REFERENCES:
- [Derived] Li C, Shoji S, Beebe J. Pharmacokinetics and C-reactive protein modelling of anti-interleukin-6 antibody (PF-04236921) in healthy volunteers and patients with autoimmune disease. Br J Clin Pharmacol. 2018 Sep;84(9):2059-2074. doi: 10.1111/bcp.13641. Epub 2018 Jun 25. PMID 29776017
- [Derived] Danese S, Vermeire S, Hellstern P, Panaccione R, Rogler G, Fraser G, Kohn A, Desreumaux P, Leong RW, Comer GM, Cataldi F, Banerjee A, Maguire MK, Li C, Rath N, Beebe J, Schreiber S. Randomised trial and open-label extension study of an anti-interleukin-6 antibody in Crohn's disease (ANDANTE I and II). Gut. 2019 Jan;68(1):40-48. doi: 10.1136/gutjnl-2017-314562. Epub 2017 Dec 15. PMID 29247068
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0151003&StudyName=A%20Study%20To%20Assess%20The%20Efficacy%20And%20Safety%20Of%20PF-04236921%20In%20Subjects%20With%20Crohn%27s%20Disease%20Who%20Failed%20Anti-TNF%20Therapy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a 28-day screening period, an induction period (Week 0-12) and a 28-week follow-up period. Participants who completed the induction treatment period could enter the follow-up period or an open-label extension study, NCT01345318. Participants who discontinued treatment during the induction period could enter the follow-up period.
Pre-assignment Details: A total of 250 participants were randomized via Interactive Voice Response System (IVRS); of which, 247 received investigational product and 3 were randomized inadvertently and not dosed (2 did not meet entrance criteria and 1 did not consent properly and was not included in clinical database because the randomization page was not completed).
Groups:
- Placebo: Placebo administered subcutaneously (SC) in the anterolateral right and left thighs on Day 1 and Day 28. Each participant received 2 injections due to the double-dummy design of the study.
- PF-04236921 10 Milligram (mg): PF-04236921 10 mg administered SC in the anterolateral right and left thighs on Day 1 and Day 28. Each participant received 2 injections due to the double-dummy design of the study.
- PF-04236921 50 mg: PF-04236921 50 mg administered SC in the anterolateral right and left thighs on Day 1 and Day 28. Each participant received 2 injections due to the double-dummy design of the study.
- PF-04236921 200 mg: PF-04236921 200 mg administered SC in the anterolateral right and left thighs on Day 1 and Day 28. Each participant received 2 injections due to the double-dummy design of the study.
Period: Overall Study
Arm/Group | Placebo | PF-04236921 10 Milligram (mg) | PF-04236921 50 mg | PF-04236921 200 mg
Started | 70 | 69 | 71 | 40 (Enrollment was halted before reaching the planned sample size due to safety findings in NCT01405196.)
Treated | 69 | 67 | 71 | 40
Completed Treatment Period | 58 | 52 | 58 | 29
Completed Follow-up Period | 3 | 8 | 3 | 4
Enrolled in NCT01345318 | 56 | 50 | 56 | 29
Completed | 59 (Include participants who completed the follow-up period or enrolled in NCT01345318.) | 58 (Include participants who completed the follow-up period or enrolled in NCT01345318.) | 59 (Include participants who completed the follow-up period or enrolled in NCT01345318.) | 33 (Include participants who completed the follow-up period or enrolled in NCT01345318.)
Not Completed | 11 | 11 | 12 | 7
Not completed — Adverse Event | 5 | 3 | 6 | 4
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 3 | 2
Not completed — Not consented properly | 0 | 1 | 0 | 0
Not completed — Not meeting entrance criteria | 1 | 1 | 0 | 0
Not completed — Other | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were summarized for the safety analysis set (SAS), which consisted of all participants who received at least 1 dose of study drug.
Groups:
- Placebo: Placebo administered SC in the anterolateral right and left thighs on Day 1 and Day 28. Each participant received 2 injections due to the double-dummy design of the study.
- PF-04236921 10 mg: PF-04236921 10 mg administered SC in the anterolateral right and left thighs on Day 1 and Day 28. Each participant received 2 injections due to the double-dummy design of the study.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg | PF-04236921 200 mg | Total
Number analyzed (Participants) | 69 | 67 | 71 | 40 | 247
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.4 (13.6) | 38.9 (12.9) | 38.9 (13.1) | 42.2 (13.2) | 39.3 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 44 | 25 | 141
  Male | 31 | 33 | 27 | 15 | 106

OUTCOME MEASURES:

1. Primary Outcome: The Crohn's Disease Activity Index (CDAI)-70 Response Rate at Week 8 in Participants Who Received Placebo, PF-04236921 10 mg and PF-04236921 50 mg
Description: CDAI-70 response was defined as a decrease in CDAI score of 70 or greater from baseline. The proportions of participants with CDAI-70 response at Week 8 were compared between placebo and PF-04236921 10 mg/50 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score greater than or equal to (>=) 0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference).
Time Frame: Baseline and Week 8
Population: Primary analysis: full analysis set (FAS, defined as all randomized participants who received at least 1 dose of study treatment; 2 participants [10 mg arm] excluded due to a quality issue) excluding 200 mg (halted prematurely before reaching the planned sample size and thus no longer powered at the planned level to test against placebo).
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg
Number analyzed (Participants) | 69 | 65 | 71
Percentage of participants | 30.6 [18.7 to 45.9] | 35.0 [21.6 to 51.1] | 49.3 [34.1 to 64.7]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 10 mg; Test type: Superiority or Other; p = 0.3406, Generalized linear mixed model (GLMM) — Type I rate was controlled for the 2 time points (Week 8 and Week 12) at 0.05 (one sided); Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 4.3, 90% CI 2-sided [-13.0 to 21.7], Standard Error of Mean 10.5
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 50 mg; Test type: Superiority or Other; p = 0.0438, GLMM — Type I rate was controlled for the 2 time points (Week 8 and Week 12) at 0.05 (one sided); Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 18.7, 90% CI 2-sided [0.7 to 36.7], Standard Error of Mean 11.0

2. Primary Outcome: The CDAI-70 Response Rate at Week 8 in Participants Who Received Placebo and PF-04236921 200 mg
Description: CDAI-70 response was defined as a decrease in CDAI score of 70 or greater from baseline. The proportions of participants with CDAI-70 response at Week 8 were compared between placebo and PF-04236921 200 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference). Since the inputs in the model included different Analysis Population than in Outcome Measure 1, that will yield different estimates for placebo for the two different models.
Time Frame: Baseline and Week 8
Population: The analysis was performed on FAS participants of the 200 mg and placebo arms, referred to as FAS 200 mg versus (vs) placebo. The 200 mg arm was halted before reaching the planned sample size of approximately 60 and was no longer powered at the planned level to test against placebo. Thus, the 200 mg vs placebo comparison is a sensitivity analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 200 mg
Number analyzed (Participants) | 69 | 40
Percentage of participants | 28.8 [15.4 to 47.4] | 39.0 [19.3 to 63.1]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 200 mg; Test type: Superiority or Other; p = 0.2258, GLMM — Type I rate was controlled for the 2 time points (Week 8 and Week 12) at 0.05 (one sided); Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 10.2, 90% CI 2-sided [-12.1 to 32.6], Standard Error of Mean 13.6

3. Primary Outcome: The CDAI-70 Response Rate at Week 12 in Participants Who Received Placebo, PF-04236921 10 mg and PF-04236921 50 mg
Description: CDAI-70 response was defined as a decrease in CDAI score of 70 or greater from baseline. The proportions of participants with CDAI-70 response at Week 12 were compared between placebo and and PF-04236921 10 mg/50 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference).
Time Frame: Baseline and Week 12
Population: Primary analysis: FAS excluding 200 mg arm (halted prematurely before reaching the planned sample size and thus no longer powered at the planned level to test against placebo).
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg
Number analyzed (Participants) | 69 | 65 | 71
Percentage of participants | 28.6 [17.1 to 43.7] | 35.2 [21.8 to 51.5] | 47.4 [32.1 to 63.1]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 10 mg; Test type: Superiority or Other; p = 0.2627, GLMM — Type I rate was controlled for the 2 time points (Week 8 and Week 12) at 0.05 (one sided); Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 6.7, 90% CI 2-sided [-10.6 to 23.9], Standard Error of Mean 10.5
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 50 mg; Test type: Superiority or Other; p = 0.0425, GLMM — Type I rate was controlled for the 2 time points (Week 8 and Week 12) at 0.05 (one sided); Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 18.8, 90% CI 2-sided [0.8 to 36.7], Standard Error of Mean 10.9

4. Primary Outcome: The CDAI-70 Response Rate at Week 12 in Participants Who Received Placebo and PF-04236921 200 mg
Description: CDAI-70 response was defined as a decrease in CDAI score of 70 or greater from baseline. The proportions of participants with CDAI-70 response at Week 12 were compared between placebo and PF-04236921 200 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference). Since the inputs in the model included different Analysis Population than in Outcome Measure 3, that will yield different estimates for placebo for the two different models.
Time Frame: Baseline and Week 12
Population: The analysis was performed on FAS 200 mg vs placebo. The 200 mg arm was halted before reaching the planned sample size of approximately 60 and was no longer powered at the planned level to test against placebo. Thus, the 200 mg vs placebo comparison is a sensitivity analysis.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 200 mg
Number analyzed (Participants) | 69 | 40
Percentage of participants | 26.7 [14.0 to 44.9] | 41.7 [21.2 to 65.6]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 200 mg; Test type: Superiority or Other; p = 0.1362, GLMM — Type I rate was controlled for the 2 time points (Week 8 and Week 12) at 0.05 (one sided); Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 15.1, 90% CI 2-sided [-7.5 to 37.6], Standard Error of Mean 13.7

5. Secondary Outcome: The CDAI-70 Response Rate Over Time in Participants Who Received Placebo, PF-04236921 10 mg and PF-04236921 50 mg
Description: CDAI-70 response was defined as a decrease in CDAI score of 70 or greater from baseline. The proportions of participants with CDAI-70 response were compared between placebo and PF-04236921 10 mg/50 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference).
Time Frame: Baseline and Weeks 2, 4, 6, and 10
Population: The analysis was performed on the FAS excluding 200 mg arm (which was halted prematurely). "n" signifies the number of subjects with observed data of each arm at each time point.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg
Number analyzed (Participants) | 69 | 65 | 71
Percentage of participants
  Week 2 (n=64, 63, 65) | 12.3 [6.3 to 22.6] | 19.4 [10.9 to 32.2] | 18.1 [10.1 to 30.3]
  Week 4 (n=66, 58, 59) | 16.5 [9.0 to 28.2] | 34.6 [21.7 to 50.3] | 37.0 [23.8 to 52.5]
  Week 6 (n=58, 53, 60) | 21.1 [11.9 to 34.6] | 35.0 [21.7 to 51.2] | 46.2 [31.6 to 61.5]
  Week 10 (n=54, 50, 51) | 29.3 [17.5 to 44.7] | 38.9 [24.4 to 55.5] | 54.0 [37.8 to 69.3]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-70 response rate for the 10-mg arm at Week 2; Test type: Superiority or Other; p = 0.1527, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 7.1, 90% CI 2-sided [-4.3 to 18.6], Standard Error of Mean 7.0
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-70 response rate for the 10-mg arm at Week 4; Test type: Superiority or Other; p = 0.0235, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 18.1, 90% CI 2-sided [3.1 to 33.2], Standard Error of Mean 9.1
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-70 response rate for the 10-mg arm at Week 6; Test type: Superiority or Other; p = 0.0792, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 13.9, 90% CI 2-sided [-2.3 to 30.2], Standard Error of Mean 9.9
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-70 response rate for the 10-mg arm at Week 10; Test type: Superiority or Other; p = 0.1909, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 9.6, 90% CI [-8.4 to 27.6], Standard Error of Mean 11.0
Statistical Analysis 5: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-70 response rate for the 50-mg arm at Week 2; Test type: Superiority or Other; p = 0.1981, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 5.8, 90% CI 2-sided [-5.4 to 17.0], Standard Error of Mean 6.8
Statistical Analysis 6: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-70 response rate for the 50-mg arm at Week 4; Test type: Superiority or Other; p = 0.0132, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 20.6, 90% CI 2-sided [5.3 to 35.8], Standard Error of Mean 9.3
Statistical Analysis 7: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-70 response rate for the 50-mg arm at Week 6; Test type: Superiority or Other; p = 0.0063, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 25.1, 90% CI 2-sided [8.6 to 41.7], Standard Error of Mean 10.1
Statistical Analysis 8: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-70 response rate for the 50-mg arm at Week 10; Test type: Superiority or Other; p = 0.0138, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 24.7, 90% CI 2-sided [6.2 to 43.1], Standard Error of Mean 11.2

6. Secondary Outcome: The CDAI-70 Response Rate Over Time in Participants Who Received Placebo and PF-04236921 200 mg
Description: CDAI-70 response was defined as a decrease in CDAI score of 70 or greater from baseline. The proportions of participants with CDAI-70 response were compared between placebo and PF-04236921 200 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference). Since the inputs in the model included different Analysis Population than in Outcome Measure 5, that will yield different estimates for placebo for the two different models.
Time Frame: Baseline and Weeks 2, 4, 6, and 10
Population: The analysis was performed on the FAS 200 mg vs placebo. The 200 mg arm was halted before reaching the planned sample size of approximately 60 participants. "n" signifies the number of subjects with observed data of each arm at each time point.
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 200 mg
Number analyzed (Participants) | 69 | 40
Percentage of participants
  Week 2 (n=64, 36) | 11.2 [5.0 to 23.1] | 26.5 [12.3 to 48.2]
  Week 4 (n=66, 35) | 15.2 [7.2 to 29.1] | 24.6 [11.2 to 45.9]
  Week 6 (n=58, 32) | 19.5 [9.6 to 35.6] | 27.2 [12.4 to 49.8]
  Week 10 (n=54, 29) | 27.2 [14.2 to 45.8] | 46.3 [24.5 to 69.7]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-70 response rate for the 200-mg arm at Week 2; Test type: Superiority or Other; p = 0.0662, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 15.4, 90% CI 2-sided [-1.4 to 32.1], Standard Error of Mean 10.2
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-70 response rate for the 200-mg arm at Week 4; Test type: Superiority or Other; p = 0.1708, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 9.5, 90% CI 2-sided [-6.9 to 25.8], Standard Error of Mean 10.0
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-70 response rate for the 200-mg arm at Week 6; Test type: Superiority or Other; p = 0.2416, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 7.8, 90% CI 2-sided [-10.5 to 26.0], Standard Error of Mean 11.1
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-70 response rate for the 200-mg arm at Week 10; Test type: Superiority or Other; p = 0.0880, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 19.1, 90% CI 2-sided [-4.1 to 42.3], Standard Error of Mean 14.1

7. Secondary Outcome: The CDAI Remission Rate Over Time in Participants Who Received Placebo, PF-04236921 10 mg and PF-04236921 50 mg
Description: CDAI remission rate was defined as an absolute CDAI score less than (<) 150. The proportions of participants with CDAI remission were compared between placebo and PF-04236921 10 mg/50 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference).
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 5
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg
Number analyzed (Participants) | 69 | 65 | 71
Percentage of participants
  Week 2 (n=64, 63, 68) | 1.6 [0.3 to 9.1] | 3.6 [1.0 to 12.3] | 9.6 [4.1 to 20.7]
  Week 4 (n=66, 58, 62) | 3.4 [0.9 to 11.6] | 4.1 [1.1 to 13.6] | 19.7 [10.0 to 35.1]
  Week 6 (n=58, 53, 63) | 8.5 [3.3 to 20.3] | 7.3 [2.6 to 19.2] | 23.4 [12.5 to 39.6]
  Week 8 (n=58, 53, 58) | 16.3 [7.6 to 31.7] | 10.8 [4.4 to 24.4] | 24.9 [13.3 to 41.7]
  Week 10 (n=54, 50, 54) | 13.1 [5.6 to 27.7] | 19.9 [9.4 to 37.2] | 30.9 [17.2 to 49.2]
  Week 12 (n=57, 52, 57) | 10.9 [4.5 to 24.1] | 10.8 [4.4 to 24.5] | 27.4 [14.9 to 44.9]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI remission rate for the 10-mg arm at Week 2; Test type: Superiority or Other; p = 0.2610, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 2.0, 90% CI 2-sided [-3.2 to 7.2], Standard Error of Mean 3.2
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI remission rate for the 10-mg arm at Week 4; Test type: Superiority or Other; p = 0.4291, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 0.7, 90% CI 2-sided [-5.6 to 7.0], Standard Error of Mean 3.8
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI remission rate for the 10-mg arm at Week 6; Test type: Superiority or Other; p = 0.5791, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = -1.2, 90% CI 2-sided [-11.0 to 8.6], Standard Error of Mean 6.0
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI remission rate for the 10-mg arm at Week 8; Test type: Superiority or Other; p = 0.7544, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = -5.5, 90% CI 2-sided [-18.8 to 7.7], Standard Error of Mean 8.0
Statistical Analysis 5: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI remission rate for the 10-mg arm at Week 10; Test type: Superiority or Other; p = 0.2308, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 6.8, 90% CI [-8.3 to 21.9], Standard Error of Mean 9.2
Statistical Analysis 6: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI remission rate for the 10-mg arm at Week 12; Test type: Superiority or Other; p = 0.5038, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = -0.1, 90% CI 2-sided [-11.8 to 11.7], Standard Error of Mean 7.1
Statistical Analysis 7: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI remission rate for the 50-mg arm at Week 2; Test type: Superiority or Other; p = 0.0498, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 8.0, 90% CI 2-sided [0.0 to 16.0], Standard Error of Mean 4.9
Statistical Analysis 8: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI remission rate for the 50-mg arm at Week 4; Test type: Superiority or Other; p = 0.0155, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 16.3, 90% CI 2-sided [3.9 to 28.7], Standard Error of Mean 7.6
Statistical Analysis 9: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI remission rate for the 50-mg arm at Week 6; Test type: Superiority or Other; p = 0.0399, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 14.9, 90% CI 2-sided [0.9 to 28.9], Standard Error of Mean 8.5
Statistical Analysis 10: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI remission rate for the 50-mg arm at Week 8; Test type: Superiority or Other; p = 0.1866, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 8.5, 90% CI 2-sided [-7.2 to 24.3], Standard Error of Mean 9.6
Statistical Analysis 11: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI remission rate for the 50-mg arm at Week 10; Test type: Superiority or Other; p = 0.0415, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 17.8, 90% CI 2-sided [0.9 to 34.7], Standard Error of Mean 10.3
Statistical Analysis 12: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI remission rate for the 50-mg arm at Week 12; Test type: Superiority or Other; p = 0.0408, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 16.5, 90% CI 2-sided [0.9 to 32.1], Standard Error of Mean 9.5

8. Secondary Outcome: The CDAI Remission Rate Over Time in Participants Who Received Placebo and PF-04236921 200 mg
Description: CDAI remission rate was defined as an absolute CDAI score <150. The proportions of participants with CDAI remission were compared between placebo and PF-04236921 200 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference). Since the inputs in the model included different Analysis Population than in Outcome Measure 7, that will yield different estimates for placebo for the two different models.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 6
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 200 mg
Number analyzed (Participants) | 69 | 40
Percentage of participants
  Week 2 (n=64, 36) | 1.1 [0.2 to 7.2] | 6.9 [1.8 to 23.1]
  Week 4 (n=66, 35) | 2.4 [0.5 to 9.8] | 5.1 [1.2 to 19.6]
  Week 6 (n=58, 32) | 6.1 [1.9 to 18.1] | 8.8 [2.4 to 27.6]
  Week 8 (n=58, 29) | 11.9 [4.3 to 29.1] | 8.8 [2.3 to 28.3]
  Week 10 (n=54, 29) | 9.4 [3.2 to 24.9] | 14.8 [4.6 to 38.5]
  Week 12 (n=57, 29) | 7.8 [2.5 to 21.5] | 11.8 [3.4 to 33.5]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI remission rate for the 200-mg arm at Week 2; Test type: Superiority or Other; p = 0.1342, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 5.8, 90% CI 2-sided [-2.8 to 14.5], Standard Error of Mean 5.3
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI remission rate for the 200-mg arm at Week 4; Test type: Superiority or Other; p = 0.2623, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 2.7, 90% CI 2-sided [-4.3 to 9.8], Standard Error of Mean 4.3
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI remission rate for the 200-mg arm at Week 6; Test type: Superiority or Other; p = 0.3324, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 2.7, 90% CI 2-sided [-7.7 to 13.2], Standard Error of Mean 6.3
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI remission rate for the 200-mg arm at Week 8; Test type: Superiority or Other; p = 0.6637, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = -3.2, 90% CI 2-sided [-15.5 to 9.1], Standard Error of Mean 7.5
Statistical Analysis 5: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI remission rate for the 200-mg arm at Week 10; Test type: Superiority or Other; p = 0.2721, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 5.4, 90% CI [-9.3 to 20.2], Standard Error of Mean 9.0
Statistical Analysis 6: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI remission rate for the 200-mg arm at Week 12; Test type: Superiority or Other; p = 0.3022, GLMM; Status of anti-TNF experience and concomitant immunosuppressant therapy were included as covariates; Mean Difference (Final Values) = 4.0, 90% CI 2-sided [-8.8 to 16.9], Standard Error of Mean 7.8

9. Secondary Outcome: The CDAI-100 Response Rate Over Time in Participants Who Received Placebo, PF-04236921 10 mg and PF-04236921 50 mg
Description: CDAI-100 response was defined as a decrease in CDAI score of 100 or greater from baseline. The proportions of participants with CDAI-100 response at Week 12 were compared between placebo and PF-04236921 10 mg/50 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference).
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 5
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg
Number analyzed (Participants) | 69 | 65 | 71
Percentage of participants
  Week 2 (n=64, 63, 65) | 12.4 [6.1 to 23.7] | 16.7 [8.8 to 29.7] | 12.6 [6.2 to 24.0]
  Week 4 (n=66, 58, 59) | 13.0 [6.5 to 24.4] | 18.1 [9.5 to 31.9] | 26.3 [15.1 to 41.8]
  Week 6 (n=58, 53, 60) | 14.5 [7.2 to 26.9] | 28.7 [16.4 to 45.1] | 32.2 [19.5 to 48.2]
  Week 8 (n=58, 53, 56) | 24.1 [13.4 to 39.3] | 26.5 [14.9 to 42.6] | 37.9 [23.7 to 54.5]
  Week 10 (n=54, 50, 51) | 21.0 [11.2 to 35.8] | 29.8 [17.0 to 46.8] | 38.2 [23.6 to 55.3]
  Week 12 (n=57, 52, 54) | 22.2 [12.1 to 37.0] | 32.7 [19.2 to 49.7] | 36.2 [22.2 to 52.9]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-100 response rate for the 10-mg arm at Week 2; Test type: Superiority or Other; p = 0.2687, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 4.3, 90% CI 2-sided [-7.2 to 15.8], Standard Error of Mean 7.0
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-100 response rate for the 10-mg arm at Week 4; Test type: Superiority or Other; p = 0.2460, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 5.1, 90% CI 2-sided [-7.1 to 17.3], Standard Error of Mean 7.4
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-100 response rate for the 10-mg arm at Week 6; Test type: Superiority or Other; p = 0.0633, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 14.2, 90% CI 2-sided [-1.1 to 29.5], Standard Error of Mean 9.3
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-100 response rate for the 10-mg arm at Week 8; Test type: Superiority or Other; p = 0.4036, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 2.4, 90% CI 2-sided [-13.8 to 18.6], Standard Error of Mean 9.9
Statistical Analysis 5: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-100 response rate for the 10-mg arm at Week 10; Test type: Superiority or Other; p = 0.1921, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 8.9, 90% CI [-7.9 to 25.6], Standard Error of Mean 10.2
Statistical Analysis 6: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in CDAI-100 response rate for the 10-mg arm at Week 12; Test type: Superiority or Other; p = 0.1541, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 10.5, 90% CI 2-sided [-6.5 to 27.5], Standard Error of Mean 10.3
Statistical Analysis 7: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-100 response rate for the 50-mg arm at Week 2; Test type: Superiority or Other; p = 0.4893, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 0.2, 90% CI 2-sided [-10.5 to 10.9], Standard Error of Mean 6.5
Statistical Analysis 8: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-100 response rate for the 50-mg arm at Week 4; Test type: Superiority or Other; p = 0.0619, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 13.2, 90% CI 2-sided [-0.9 to 27.4], Standard Error of Mean 8.6
Statistical Analysis 9: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-100 response rate for the 50-mg arm at Week 6; Test type: Superiority or Other; p = 0.0290, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 17.7, 90% CI 2-sided [2.3 to 33.1], Standard Error of Mean 9.3
Statistical Analysis 10: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-100 response rate for the 50-mg arm at Week 8; Test type: Superiority or Other; p = 0.0988, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 13.8, 90% CI 2-sided [-3.8 to 31.4], Standard Error of Mean 10.7
Statistical Analysis 11: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-100 response rate for the 50-mg arm at Week 10; Test type: Superiority or Other; p = 0.0549, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 17.2, 90% CI 2-sided [-0.5 to 35.0], Standard Error of Mean 10.8
Statistical Analysis 12: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in CDAI-100 response rate for the 50-mg arm at Week 12; Test type: Superiority or Other; p = 0.0920, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 14.0, 90% CI 2-sided [-3.3 to 31.3], Standard Error of Mean 10.5

10. Secondary Outcome: The CDAI-100 Response Rate Over Time in Participants Who Received Placebo and PF-04236921 200 mg
Description: CDAI-100 response was defined as a decrease in CDAI score of 100 or greater from baseline. The proportions of participants with CDAI-100 response at Week 12 were compared between placebo and PF-04236921 200 mg. CDAI is used to quantify the symptoms of patients with Crohn's Disease. CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit. Many clinical trials use the endpoint for response as a 70 or greater point decrease in CDAI and clinical remission is often defined as a CDAI score below 150. The Outcome included a Generalized linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference). Since the inputs in the model included different Analysis Population than in Outcome Measure 9, that will yield different estimates for placebo for the two different models.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 6
Measure: Least Squares Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | PF-04236921 200 mg
Number analyzed (Participants) | 69 | 40
Percentage of participants
  Week 2 (n=64, 36) | 10.3 [4.4 to 22.6] | 12.0 [4.5 to 28.6]
  Week 4 (n=66, 35) | 11.0 [4.7 to 23.5] | 22.1 [9.5 to 43.5]
  Week 6 (n=58, 32) | 12.2 [5.3 to 25.8] | 22.2 [9.3 to 44.2]
  Week 8 (n=58, 29) | 21.3 [10.3 to 39.1] | 18.7 [7.3 to 40.2]
  Week 10 (n=54, 29) | 18.2 [8.4 to 34.9] | 30.4 [13.6 to 54.8]
  Week 12 (n=57, 29) | 19.4 [9.2 to 36.5] | 26.9 [11.6 to 50.6]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-100 response rate for the 200-mg arm at Week 2; Test type: Superiority or Other; p = 0.4031, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 1.7, 90% CI 2-sided [-9.5 to 12.9], Standard Error of Mean 6.8
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-100 response rate for the 200-mg arm at Week 4; Test type: Superiority or Other; p = 0.1219, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 11.1, 90% CI 2-sided [-4.6 to 26.8], Standard Error of Mean 9.6
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-100 response rate for the 200-mg arm at Week 6; Test type: Superiority or Other; p = 0.1600, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 9.9, 90% CI 2-sided [-6.5 to 26.4], Standard Error of Mean 10.0
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-100 response rate for the 200-mg arm at Week 8; Test type: Superiority or Other; p = 0.6019, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -2.7, 90% CI 2-sided [-19.5 to 14.2], Standard Error of Mean 10.3
Statistical Analysis 5: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-100 response rate for the 200-mg arm at Week 10; Test type: Superiority or Other; p = 0.1601, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 12.3, 90% CI [-8.0 to 32.5], Standard Error of Mean 12.3
Statistical Analysis 6: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in CDAI-100 response rate for the 200-mg arm at Week 12; Test type: Superiority or Other; p = 0.2622, GLMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 7.4, 90% CI 2-sided [-11.8 to 26.6], Standard Error of Mean 11.7

11. Secondary Outcome: Change From Baseline in CDAI Score Over Time in Participants Who Received Placebo, PF-04236921 10 mg and PF-04236921 50 mg
Description: CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit, and higher score indicate more severe disease. The Outcome included a Linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference).
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 5
Measure: Least Squares Mean (90% Confidence Interval); unit: points on a scale
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg
Number analyzed (Participants) | 69 | 65 | 71
points on a scale
  Week 2 (n=64, 63, 65) | -18.9 [-38.3 to 0.6] | -28.4 [-47.6 to -9.3] | -16.2 [-34.5 to 2.2]
  Week 4 (n=66, 58, 59) | -25.1 [-44.9 to -5.2] | -37.1 [-57.0 to -17.1] | -50.7 [-70.0 to -31.5]
  Week 6 (n=58, 53, 60) | -32.6 [-55.5 to -9.6] | -48.5 [-71.7 to -25.3] | -54.9 [-77.0 to -32.9]
  Week 8 (n=58, 53, 56) | -34.6 [-58.8 to -10.5] | -49.6 [-74.1 to -25.0] | -63.5 [-86.9 to -40.0]
  Week 10 (n=54, 50, 51) | -19.8 [-45.9 to 6.4] | -50.0 [-76.6 to -23.4] | -64.7 [-90.3 to -39.1]
  Week 12 (n=57, 52, 54) | -27.3 [-53.5 to -1.2] | -44.2 [-70.9 to -17.5] | -66.8 [-92.5 to -41.2]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in change from baseline in CDAI score for the 10-mg arm at Week 2; Test type: Superiority or Other; p = 0.2173, Linear mixed model (LMM); Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -9.6, 90% CI 2-sided [-29.8 to 10.6], Standard Error of Mean 12.22
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in change from baseline in CDAI score for the 10-mg arm at Week 4; Test type: Superiority or Other; p = 0.1778, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -12.0, 90% CI 2-sided [-33.4 to 9.4], Standard Error of Mean 12.95
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in change from baseline in CDAI score for the 10-mg arm at Week 6; Test type: Superiority or Other; p = 0.1661, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -15.9, 90% CI 2-sided [-43.0 to 11.2], Standard Error of Mean 16.37
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in change from baseline in CDAI score for the 10-mg arm at Week 8; Test type: Superiority or Other; p = 0.1993, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -14.9, 90% CI 2-sided [-44.1 to 14.3], Standard Error of Mean 17.66
Statistical Analysis 5: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in change from baseline in CDAI score for the 10-mg arm at Week 10; Test type: Superiority or Other; p = 0.0632, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -30.2, 90% CI 2-sided [-62.7 to 2.3], Standard Error of Mean 19.66
Statistical Analysis 6: Comparison: Placebo vs PF-04236921 10 mg; LSM difference from placebo in change from baseline in CDAI score for the 10-mg arm at Week 12; Test type: Superiority or Other; p = 0.1975, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -16.8, 90% CI 2-sided [-49.4 to 15.8], Standard Error of Mean 19.71
Statistical Analysis 7: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in change from baseline in CDAI score for the 50-mg arm at Week 2; Test type: Superiority or Other; p = 0.5868, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = 2.7, 90% CI 2-sided [-17.6 to 22.9], Standard Error of Mean 12.25
Statistical Analysis 8: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in change from baseline in CDAI score for the 50-mg arm at Week 4; Test type: Superiority or Other; p = 0.0243, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -25.7, 90% CI 2-sided [-47.0 to -4.3], Standard Error of Mean 12.93
Statistical Analysis 9: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in change from baseline in CDAI score for the 50-mg arm at Week 6; Test type: Superiority or Other; p = 0.0834, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -22.4, 90% CI 2-sided [-49.0 to 4.3], Standard Error of Mean 16.12
Statistical Analysis 10: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in change from baseline in CDAI score for the 50-mg arm at Week 8; Test type: Superiority or Other; p = 0.0499, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -28.8, 90% CI 2-sided [-57.7 to -0.0], Standard Error of Mean 17.43
Statistical Analysis 11: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in change from baseline in CDAI score for the 50-mg arm at Week 10; Test type: Superiority or Other; p = 0.0111, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -44.9, 90% CI 2-sided [-77.1 to -12.7], Standard Error of Mean 19.45
Statistical Analysis 12: Comparison: Placebo vs PF-04236921 50 mg; LSM difference from placebo in change from baseline in CDAI score for the 50-mg arm at Week 12; Test type: Superiority or Other; p = 0.0221, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -39.5, 90% CI 2-sided [-71.7 to -7.3], Standard Error of Mean 19.49

12. Secondary Outcome: Change From Baseline in CDAI Score Over Time in Participants Who Received Placebo and PF-04236921 200 mg
Description: CDAI evaluates 8 Crohn's disease-related variables during a 1-week assessment period, yielding a composite score >=0 and without an upper limit, and higher score indicate more severe disease. The Outcome included a Linear mixed model analyses which incorporated longitudinal data for each subject, and the same model is used for estimate (least squares mean) and statistical analysis (mean difference). Since the inputs in the model included different Analysis Population than in Outcome Measure 11, that will yield different estimates for placebo for the two different models.
Time Frame: Baseline and Weeks 2, 4, 6, 8, 10, and 12
Population: as for outcome 6
Measure: Least Squares Mean (90% Confidence Interval); unit: points on a scale
Arm/Group | Placebo | PF-04236921 200 mg
Number analyzed (Participants) | 69 | 40
points on a scale
  Week 2 (n=64, 36) | -21.3 [-49.1 to 6.6] | -30.1 [-62.2 to 2.1]
  Week 4 (n=66, 35) | -26.6 [-54.3 to 1.1] | -30.5 [-62.5 to 1.6]
  Week 6 (n=58, 32) | -36.7 [-64.6 to -8.7] | -42.2 [-74.8 to -9.6]
  Week 8 (n=58, 29) | -39.1 [-67.2 to -11.0] | -48.1 [-81.3 to -14.9]
  Week 10 (n=54, 29) | -26.3 [-54.7 to 2.1] | -56.1 [-89.5 to -22.7]
  Week 12 (n=57, 29) | -35.2 [-63.6 to -6.8] | -66.2 [-99.9 to -32.6]
Statistical Analysis 1: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in change from baseline in CDAI score for the 200-mg arm at Week 2; Test type: Superiority or Other; p = 0.3157, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -8.8, 90% CI 2-sided [-39.0 to 21.4], Standard Error of Mean 18.27
Statistical Analysis 2: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in change from baseline in CDAI score for the 200-mg arm at Week 4; Test type: Superiority or Other; p = 0.4171, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -3.8, 90% CI 2-sided [-34.0 to 26.4], Standard Error of Mean 18.28
Statistical Analysis 3: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in change from baseline in CDAI score for the 200-mg arm at Week 6; Test type: Superiority or Other; p = 0.3837, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -5.6, 90% CI 2-sided [-36.6 to 25.5], Standard Error of Mean 18.79
Statistical Analysis 4: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in change from baseline in CDAI score for the 200-mg arm at Week 8; Test type: Superiority or Other; p = 0.3204, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -9.0, 90% CI 2-sided [-40.8 to 22.8], Standard Error of Mean 19.27
Statistical Analysis 5: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in change from baseline in CDAI score for the 200-mg arm at Week 10; Test type: Superiority or Other; p = 0.0649, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -29.9, 90% CI 2-sided [-62.3 to 2.6], Standard Error of Mean 19.64
Statistical Analysis 6: Comparison: Placebo vs PF-04236921 200 mg; LSM difference from placebo in change from baseline in CDAI score for the 200-mg arm at Week 12; Test type: Superiority or Other; p = 0.0598, LMM; Status of anti-TNF experience, concomitant immunosuppressant therapy, and baseline were included as covariates; Mean Difference (Final Values) = -31.0, 90% CI 2-sided [-63.9 to 1.8], Standard Error of Mean 19.87

13. Secondary Outcome: Percentages of Participants With Confirmed Positive Anti-drug Antibodies (ADAs)
Description: The percentage of participants with confirmed positive ADA was summarized for each treatment arm. ADA positive was defined as ADA titer defined as ADA titer (ie, the reciprocal of the highest dilution that gives a value equivalent to the cut point of the assay) >= 4.32.
Time Frame: At baseline (Day 1) and at Weeks 4, 8, 12, 16, 24, 32 and 40
Population: The SAS consisted of all participants who received at least 1 dose of study drug. "n" signifies number of participants with observed data at the time point of each arm. From Weeks 16 to 40, only participants who remained in the follow-up period of this study and did not enter NCT01405196 were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04236921 10 mg | PF-04236921 50 mg | PF-04236921 200 mg
Number analyzed (Participants) | 67 | 71 | 40
percentage of participants
  Day 1 (n=56, 66, 36) | 0.0 | 0.0 | 0.0
  Week 4 (n=58, 62, 29) | 0.0 | 1.6 | 0.0
  Week 8 (n=53, 53, 27) | 0.0 | 0.0 | 0.0
  Week 12 (n=46, 49, 24) | 0.0 | 0.0 | 0.0
  Week 16 (n=2, 1, 0) | 0.0 | 0.0 | NA — No participants analyzed.
  Week 24 (n=2, 1, 0) | 0.0 | 0.0 | NA — No participants analyzed.
  Week 32 (n=1, 0, 0) | 0.0 | NA — No participants analyzed. | NA — No participants analyzed.
  Week 40 (n=2, 1, 0) | 0.0 | 0.0 | NA — No participants analyzed.

14. Secondary Outcome: Percentages of Participants With Confirmed Positive Neutralizing Antibodies (NAbs)
Description: The percentage of participants with confirmed positive NAbs was summarized for each treatment arm. Only ADA positive samples were analyzed for Nab. A multi-tiered approach was utilized to detect NAbs. NAb serum samples were screened at tier one, and those found presumptively NAb positive was further tested with the confirmatory assay (tier two). The percentage of subjects with confirmed positive NAbs was summarized for each treatment.
Time Frame: At baseline (Day 1) and at Weeks 4, 8, 12, 16, 24, 32 and 40
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | PF-04236921 10 mg | PF-04236921 50 mg | PF-04236921 200 mg
Number analyzed (Participants) | 67 | 71 | 40
percentage of participants
  Day 1 (n=56, 66, 36) | 0.0 | 0.0 | 0.0
  Week 4 (n=58, 62, 29) | 0.0 | 1.6 | 0.0
  Week 8 (n=53, 53, 27) | 0.0 | 0.0 | 0.0
  Week 12 (n=46, 49, 24) | 0.0 | 0.0 | 0.0
  Week 16 (n=2, 1, 0) | 0.0 | 0.0 | NA — No participants analyzed.
  Week 24 (n=2, 1, 0) | 0.0 | 0.0 | NA — No participants analyzed.
  Week 32 (n=1, 0, 0) | 0.0 | NA — No participants analyzed. | NA — No participants analyzed.
  Week 40 (n=2, 1, 0) | 0.0 | 0.0 | NA — No participants analyzed.

15. Secondary Outcome: Serum PF-04236921 Concentration Over Time
Time Frame: Day 1 (predose), and at Weeks 2, 4 (Day 28, predose), 8, 10, 12, 16, 20, 24, 28, 32, 36, and 40
Population: The pharmacokinetic (PK) analysis set was the subset of participants from the SAS who provided at least 1 PK concentration (2 participants [10 mg arm] excluded due to a quality issue). "n" is the number of participants with PK data at the visit. From Weeks 16 to 40, only participants who remained in the follow-up period of this study were analyzed.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-04236921 10 mg | PF-04236921 50 mg | PF-04236921 200 mg
Number analyzed (Participants) | 65 | 71 | 40
nanogram per milliliter (ng/mL)
  Day 1 (n=54, 64, 37) | 4.52 (33.20) | 2.05 (16.38) | NA (NA) — Concentrations were not determined due to being below the lower limit of quantification (<LLOQ)
  Week 2 (n=46, 56, 30) | 1060 (531.3) | 4580 (1938) | 21300 (9547)
  Week 4 (n=56, 63, 29) | 674 (339.3) | 3180 (1555) | 14800 (6641)
  Week 6 (n=48, 57, 28) | 1470 (863.0) | 6610 (2668) | 32200 (13240)
  Week 8 (n=51, 52, 28) | 992 (501.7) | 4500 (1993) | 20200 (8683)
  Week 10 (n=47, 54, 29) | 695 (428.5) | 3280 (1961) | 13600 (7350)
  Week 12 (n=43, 51, 26) | 504 (435.5) | 2110 (1333) | 10900 (7802)
  Week 16 (n=2, 1, 0) | 177 (250.3) | 1290 (NA) — Standard deviation was not calculable as there was only 1 participant. | NA (NA) — Number of participants analyzed was 0 at the visit
  Week 20 (n=2, 1, 0) | 102 (143.5) | 425 (NA) — Standard deviation was not calculable as there was only 1 participant. | NA (NA) — Number of participants analyzed was 0 at the visit
  Week 24 (n=2, 1, 0) | 63.5 (89.80) | NA (NA) — Concentrations were not determined due to <LLOQ | NA (NA) — Number of participants analyzed was 0 at the visit
  Week 28 (n=2, 0, 0) | NA (NA) — Concentrations were not determined due to <LLOQ | NA (NA) — Number of participants analyzed was 0 at the visit | NA (NA) — Number of participants analyzed was 0 at the visit
  Week 32 (n=2, 0, 0) | NA (NA) — Concentrations were not determined due to <LLOQ | NA (NA) — Number of participants analyzed was 0 at the visit | NA (NA) — Number of participants analyzed was 0 at the visit
  Week 36 (n=2, 1, 0) | NA (NA) — Concentrations were not determined due to <LLOQ | 109 (NA) — Standard deviation was not calculable as there was only 1 participant. | NA (NA) — Number of participants analyzed was 0 at the visit
  Week 40 (n=2, 1, 0) | NA (NA) — Concentrations were not determined due to <LLOQ | NA (NA) — Concentrations were not determined due to <LLOQ | NA (NA) — Number of participants analyzed was 0 at the visit

16. Secondary Outcome: Number of Participants Who Withdrew From the Study Due to Treatment-emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. Treatment-emergent were events between first dose of treatment and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Induction period: from Week 0 (Day 1) through Week 12; follow-up period: from Week 12 (or discontinuation from the induction period) through last subject visit (up to 28 weeks after completion of or discontinuation from the 12-week induction period)
Population: as for outcome 13
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg | PF-04236921 200 mg
Number analyzed (Participants) | 69 | 67 | 71 | 40
participants
  Induction period (Weeks 0 to 12) | 7 | 6 | 6 | 8
  Follow-up period (after Week 12) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The reporting period was from the time of the first dose of study treatment through last subject visit up to 40 weeks post the first dose of study treatment for serious adverse events (SAEs) and other adverse events (AEs).
Description: The same event may appear as both an AE and an SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | Placebo | PF-04236921 10 mg | PF-04236921 50 mg | PF-04236921 200 mg
Serious Adverse Events (participants affected / at risk) | 11/69 | 11/67 | 12/71 | 11/40
Other Adverse Events (participants affected / at risk) | 36/69 | 38/67 | 48/71 | 20/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=69) | PF-04236921 10 mg (N=67) | PF-04236921 50 mg (N=71) | PF-04236921 200 mg (N=40)
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 6 | 6 | 5 | 4
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 2 | 0
Groin abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Retroperitoneal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=69) | PF-04236921 10 mg (N=67) | PF-04236921 50 mg (N=71) | PF-04236921 200 mg (N=40)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 6 | 8 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Crohn's disease (Gastrointestinal disorders) | 4 | 2 | 7 | 4
Nausea (Gastrointestinal disorders) | 1 | 8 | 7 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 2 | 5 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 5 | 2
Fatigue (General disorders) | 0 | 2 | 4 | 0
Pyrexia (General disorders) | 7 | 5 | 5 | 1
Nasopharyngitis (Infections and infestations) | 3 | 11 | 8 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 4 | 0
Urinary tract infection (Infections and infestations) | 3 | 4 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 5 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 1
Headache (Nervous system disorders) | 6 | 4 | 9 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 7 | 1

LIMITATIONS AND CAVEATS:
Enrollment into the 200 mg arm was halted on 14 August 2013 before reaching the planned sample size due to safety findings in NCT01405196. Hence the 200 mg vs placebo comparisons were excluded from the primary analyses and reported separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigators will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.